CLINICAL TRIAL: NCT03377426
Title: A Randomized, Controlled, Evaluator-blinded, Multi-center, Study to Evaluate LYS228 Pharmacokinetics, Clinical Response, Safety and Tolerability in Patients With Complicated Urinary Tract Infection
Brief Title: LYS228 PK, Clinical Response, Safety and Tolerability in Patients With Complicated Urinary Tract Infection (cUTI)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated due to an out-licensing agreement after the new sponsor did not wish to continue the trial
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CLYS228X2201
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Complicated Urinary Tract Infections
Keywords: Urinary tract infection, LYS228, beta-lactam antibiotics, creatinine clearance, Enterobactericeae
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded evaluator will perform the safety and efficacy assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYS228 (Experimental): IV infusion
  Interventions: Drug: LYS228
- Standard of care (Active Comparator): IV infusion of standard of care antibiotics for at least 5 days
  Interventions: Drug: Standard of care therapy

INTERVENTIONS:
Drug: LYS228 — LYS228 IV infusion
  Arms: LYS228
Drug: Standard of care therapy — IV infusion of standard of care antibiotics
  Arms: Standard of care

SUMMARY:
The purpose of the study is to evaluate whether LYS228 can be developed for the treatment of complicated urinary tract infections

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 85 years of age with suspected and/or bacteriologically documented complicated UTI judges by the investigator to be serious (required patient to be hospitalized for treatment with intravenous antibiotics)

Exclusion Criteria:

* Urine Gram stain that demonstrated that a Gram-positive organism was present, or if urine culture results were available, demonstrated Gram- positive organisms were present at ≥10E5 CFU/mL
* Urine culture result available at enrollment and demonstrating more than 2 different species of microorganisms regardless of the colony count
* Urine culture result available demonstrating fungal UTI with colony count >10E3 CFU/mL
* Patient had received prior antibiotics within 72 hours before the initiation of study therapy
* Patients with estimated glomerular filtration rate < 30mL/min calculated based in study qualified formula

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-19 (Estimated); Primary Completion 2019-10-28 (Estimated); Study Completion 2019-10-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of the Clinical Response at Day 7 | Baseline, Day 7
  Clinical success at 7 days after randomization determined by signs and symptoms of infection and the need for additional antibiotics
Plasma Pharmacokinetics (PK) of LYS228: Area Under the Plasma Concentration-time Curve from time zero to the end of dosing interval tau (AUCtau) | Day 5
  Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Plasma Pharmacokinetics (PK) of LYS228: The observed maximum plasma concentration following drug administration (Cmax) | Day 5
  Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Plasma Pharmacokinetics (PK) of LYS228: The time to reach the maximum concentration after drug administration (Tmax) | Day 5
  Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Plasma Pharmacokinetics (PK) of LYS228: The systemic (or total body) clearance from plasma following intravenous administration (CL) | Day 5
  Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Plasma Pharmacokinetics (PK) of LYS228: The volume of distribution at steady state following intravenous administration (Vss) | Day 5
  Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Plasma Pharmacokinetics (PK) of LYS228: The terminal elimination half-life (T 1/2) | Day 5
  Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Plasma Pharmacokinetics (PK) of LYS228: The amount of time in which the unbound drug concentration exceeds the minimum inhibitory concentration of the organism (%fT>MIC) | Day 5
  Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Urine Pharmacokinetics (PK) of LYS228: The amount of drug eliminated in Urine from 0 hours up to 6 hours following intravenus administration (Ae0-6h) | Day 5
  Calculated based on LYS228 concentration in urine at different time points following drug administration on Day 5
Urine Pharmacokinetics (PK) of LYS228: Renal Clearance (CLr) | Day 5
  Calculated based on LYS228 concentration in urine at different time points following drug administration on Day 5

SECONDARY OUTCOMES:
Change from Baseline of the Microbiological Response at Day 7 | Baseline, Day 7
  Microbiologic success at 7 days after randomization determined by microbial growth in urine culture

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Seattle, Washington
- Novartis Investigative Site, Odense, Denmark
- Novartis Investigative Site, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Dean CR, Barkan DT, Bermingham A, Blais J, Casey F, Casarez A, Colvin R, Fuller J, Jones AK, Li C, Lopez S, Metzger LE 4th, Mostafavi M, Prathapam R, Rasper D, Reck F, Ruzin A, Shaul J, Shen X, Simmons RL, Skewes-Cox P, Takeoka KT, Tamrakar P, Uehara T, Wei JR. Mode of Action of the Monobactam LYS228 and Mechanisms Decreasing In Vitro Susceptibility in Escherichia coli and Klebsiella pneumoniae. Antimicrob Agents Chemother. 2018 Sep 24;62(10):e01200-18. doi: 10.1128/AAC.01200-18. Print 2018 Oct. PMID 30061293